CLINICAL TRIAL: NCT04205162
Title: Evaluating the Initial Lens Handling Experience of Neophyte Contact Lens Wearers Fitted With Precision1 and 1-Day Acuvue Moist Contact Lenses
Acronym: SALUKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41693
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators will be masked to which lens type (brand) the participants will be wearing in each eye during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Verofilcon A / Etafilcon A (Experimental): The participant will wear Verofilcon A in their right eye and Etafilcon A in their left eye.
  Interventions: Device: Verafilcon A; Device: Etafilcon A
- Etafilcon A / Verofilcon A (Experimental): The participant will wear Etafilcon A in their right eye and Verafilcon A in their left eye.
  Interventions: Device: Verafilcon A; Device: Etafilcon A

INTERVENTIONS:
Device: Verafilcon A — Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Other Names: Precision1™
Device: Etafilcon A — Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Other Names: Acuvue® Moist

SUMMARY:
The initial subjecting handling experience of neophyte contact lens wearers with Precision1 will be compared to that with a daily disposable lens which mas been on the market for numerous years (1-Day ACUVUE Moist).

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 40 years of age inclusively and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is a neophyte who has no history of any previous contact lens handling experience;
5. Has a refraction cyl ≤1.00DC in either eye (after vertexing to corneal plane);
6. Has visual acuity ≤0.20 logMAR each eye with study lenses;
7. Demonstrates acceptable fit with study lenses;
8. Demonstrates the ability to successfully insert and remove the study lenses 3 times for each eye (contralateral CL handling, so that each lens type inserted and removed 3x on same eye);
9. Is willing to wear study CLs at least 5 days per week and 6 hours per day throughout the study

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by self-report);
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has taken part in another clinical research study within the last 14 days;
10. Any ocular and/or systemic conditions or concomitant medication to contraindicate contact lens wear or be expected to interfere with the primary outcome variables.

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between December 2019 and May 2022. The first participant was enrolled on December 13, 2019 and the last participant was enrolled on May 20, 2022.
Pre-assignment Details: Of 40 enrolled participants, 36 met inclusion criteria and were randomized to treatment.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Verofilcon A / Etafilcon A | Etafilcon A / Verofilcon A
Started | 18; 36 eyes | 18; 36 eyes
Completed | 14; 28 eyes | 18; 36 eyes
Not Completed | 4; 8 eyes | 0; 0 eyes
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — University closure due to COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verofilcon A / Etafilcon A | Etafilcon A / Verofilcon A | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.3 (3.3) | 23.7 (4.0) | 23.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings of Lens Handling for Insertion Per Intervention
Description: At the initial visit, once participants had successfully completed contact lens insertion and removal training, participants were asked to rate the subjective handling of the lens for insertion on a scale from 0 (worst) to 100 (best) using a visual analog scale per intervention. Higher scores indicate that the lens was very easy to insert.
Time Frame: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Verofilcon A / Etafilcon A | Etafilcon A / Verofilcon A
Number analyzed (Participants) | 18 | 18
score on a scale
  verofilcon A | 85 [50 to 99] | 80 [17 to 95]
  etafilcon A | 75 [10 to 100] | 85 [50 to 99]
Statistical Analysis 1: Comparison: Verofilcon A / Etafilcon A vs Etafilcon A / Verofilcon A; Comparison of etafilcon A; Test type: Other; p = 0.331, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Verofilcon A / Etafilcon A vs Etafilcon A / Verofilcon A; Comparison of verofilcon A; Test type: Other; p = 0.122, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Subjective Ratings of Lens Handling for Removal Per Intervention
Description: At the initial visit, once participants had successfully completed contact lens insertion and removal training, participants were asked to rate the subjective handling of the lens for removal on a scale from 0 (worst) to 100 (best) using a visual analog scale per intervention. Higher scores indicate that the lens was very easy to remove.
Time Frame: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Verofilcon A / Etafilcon A | Etafilcon A / Verofilcon A
Number analyzed (Participants) | 18 | 18
score on a scale
  etaflicon A | 80 [30 to 100] | 90 [25 to 99]
  verofilcon A | 70 [20 to 95] | 72.50 [25 to 95]
Statistical Analysis 1: Comparison: Verofilcon A / Etafilcon A vs Etafilcon A / Verofilcon A; Comparison of etafilcon A; Test type: Other; p = 0.130, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Verofilcon A / Etafilcon A vs Etafilcon A / Verofilcon A; Comparison of verofilcon A; Test type: Other; p = 0.924, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Average of 1 week
Description: An adverse event was defined as any unfavourable and unintended sign, symptom, or disease temporarily associated with a study procedure, whether there was a causal relationship or not.
Groups:
- Ocular Adverse Events Only: Verofilcon A (Per Intervention): The participant will wear Verofilcon A in one eye.
  Verafilcon A: Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Ocular adverse events are reported per intervention.
- Ocular Adverse Events Only: Etafilcon A (Per Intervention): The participant will wear Etafilcon A in the other eye.
  Etafilcon A: Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Ocular adverse events are reported per intervention.
- Systemic Adverse Events: Verofilcon A and Etafilcon A: The participant will wear Verofilcon A in one eye and Etafilcon A in the other eye.
  Verafilcon A: Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Etafilcon A: Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
Arm/Group | Ocular Adverse Events Only: Verofilcon A (Per Intervention) | Ocular Adverse Events Only: Etafilcon A (Per Intervention) | Systemic Adverse Events: Verofilcon A and Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 1/36 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocular Adverse Events Only: Verofilcon A (Per Intervention) (N=36) | Ocular Adverse Events Only: Etafilcon A (Per Intervention) (N=36) | Systemic Adverse Events: Verofilcon A and Etafilcon A (N=36)
Ocular irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Ocular irritation due to lens wear. Mild increase in redness.
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was affected by the COVID-19 pandemic, which resulted in a mandated site closure to limit the spread of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT04205162/Prot_SAP_000.pdf